CLINICAL TRIAL: NCT00942006
Title: Doxycycline and Ceftriaxone in Patients With Suspected Early Lyme Neuroborreliosis and Normal CSF Cell Count.
Brief Title: Doxycycline and Ceftriaxone in Suspected Early Lyme Neuroborreliosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Katarina Ogrinc MD PhD, UMC Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LNB-doxy-ceftriaxone
Record Dates: First submitted 2009-07-17; First posted 2009-07-20 (Estimated); Last update posted 2009-07-20 (Estimated); Status verified 2009-07

CONDITIONS: Suspected Early Lyme Neuroborreliosis
Keywords: Lyme neuroborreliosis; Lyme borreliosis; erythema migrans; doxycycline treatment; ceftriaxone treatment; outcome; subjective symptoms
MeSH Terms: conditions — Lyme Neuroborreliosis; Lyme Disease; Glossitis, Benign Migratory | interventions — Doxycycline; Ceftriaxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LNB-doxycycline (Active Comparator)
  Interventions: Drug: doxycycline
- LNB-ceftriaxone (Active Comparator)
  Interventions: Drug: ceftriaxone

INTERVENTIONS:
Drug: doxycycline — 100 mg bid, 14 days
  Arms: LNB-doxycycline
Drug: ceftriaxone — 2g x 1 iv, 14 days
  Arms: LNB-ceftriaxone

SUMMARY:
The investigators will compare doxycycline and ceftriaxone in treatment of patients with suspected early Lyme neuroborreliosis and normal CSF cell count. The study hypothesis is that the efficacy and adverse effects of both antibiotics are comparable.

ELIGIBILITY:
Inclusion Criteria:

* age >15 years
* erythema migrans in 4 months period before neurologic symptoms
* normal CSF cell count
* absence of more defined clinical symptoms or signs for CNS involvement (radicular pain, meningeal signs, peripheral facial palsy).

Exclusion Criteria:

* pregnancy
* lactation
* allergy on doxycycline and ceftriaxone
* immune deficiency.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Objective sequelae and post-treatment subjective symptoms in patients treated for suspected early Lyme neuroborreliosis with normal CSF cell count with doxycycline or ceftriaxone for 14 days. | 1 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Franc Strle, MD PhD, Study Chair — UMC Ljubljana
Locations (1):
- UMC Ljubljana, Department of Infectious Diseases, Ljubljana, Slovenia